CLINICAL TRIAL: NCT05919394
Title: Increase in Inhaled Corticosteroid Dose vs Triple Therapy in T2-high Asthma Patients Who Remain Uncontrolled With Medium Dose Inhaled Corticosteroids/Long-acting β2 Adrenergic Combination: a Real-life Study. TRICORDA Study
Brief Title: Triple vs High Dose Inhaled CORticosteroids
Acronym: TRICORDA
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study is closed due to lack of recruitment.
Sponsor: Galaxia Empírica (Network)
Collaborators: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRICORDA
Record Dates: First submitted 2023-06-01; First posted 2023-06-26 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Asthma
Keywords: Wheezing; Dyspnoea; Cough
MeSH Terms: conditions — Asthma; Respiratory Sounds; Dyspnea; Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Triple treatment with medium doses of CSI/LABA/LA (Active Comparator): Medium-dose inhaled triple therapy of inhaled corticosteroid: IC, long-acting beta-agonist: LABA and anticholinergic: LAMA
  Interventions: Drug: To compare in both treatment arms the percentage of patients controlled at week 52.
- Treatment with high doses of CSI/LABA (Active Comparator): High doses of of inhaled corticosteroid: IC and long-acting beta-agonist: LABA
  Interventions: Drug: To compare in both treatment arms the percentage of patients controlled at week 52.

INTERVENTIONS:
Drug: To compare in both treatment arms the percentage of patients controlled at week 52. — Participants will be assigned to receive one of two therapeutic strategies: the same ICS/LABA combination at the higher doses or the same maintenance treatment at medium doses plus a LAMA.
  Other Names: Triple therapy

SUMMARY:
Increase in inhaled corticosteroid dose vs triple therapy in T2-high asthma patients who remain uncontrolled with medium dose inhaled corticosteroids/long-acting β2 adrenergic combination: a real-life study.

DETAILED DESCRIPTION:
It remains to be clarified whether triple therapy is better than high dose inhaled corticosteroids and long-acting beta2-agonists combination (ICS/LABA) in patients with uncontrolled asthma despite the use of medium dose ICS/LABA combinations, particularly in cases with high T2 biomarkers´ values. The aim of this study is to evaluate, in a real-world setting, which is the best therapeutic strategy in this clinical scenario.

This study will be a randomized, open-label, two-arm, prospective, 12-month trial to be conducted in 53 hospital asthma units. Participants will be allocated to receive one of two therapeutic strategies: same ICS/LABA combination at highest doses or the same maintenance therapy plus a long-acting anticholinergic (LAMA). Follow up visits will be scheduled at 12-16, 24-28 and 52 weeks after the baseline visit. The investigators can optimise therapy according to their clinical opinion if the patient remains uncontrolled. Demographic, clinical and lung function information will be collected at each visit.

The primary endpoint will be the percentage of patients controlled at week 52, with both an ACT score of 20 or greater and no severe exacerbations). 620 patients (282 patients per treatment group, considering 10% drop-out) will be required for the study to have 80% power to detect non-inferiority limit of 10% in the rate of controlled patients between the high dose ICS/LABA arm and the triple therapy arm. All effectiveness analyses will be done according to the intention-to-treat principle. Secondary endpoints: percentage of patients controlled at week 24, ACT at weeks 12, 24 and 52, AIRQ at weeks 12, 24 and 52, quality of life (Mini-AQLQ) at weeks 12, 24 and 52, postbronchodilator FEV1 at weeks 12, 24 and 52, severe exacerbations at week 24 and 52. Differences between groups in 8 AM serum cortisol at week 52. Adherence at week 52 in the two study arms. Factors related to triple and high-dose ICS/LABA failure and success (control) at week 52.

The results of this study will help physicians to decide the most appropriate therapeutic strategy for a large number of asthma patients: those who do not gain control with medium dose ICS/LABA. If non-inferiority of triple therapy vs high dose ICS/LABA is demonstrated, it could lead to a modification of the current guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 80 years of age diagnosed of uncontrolled asthma.
* T2 high asthma: > 300 cels/mm3 blood Eos (current value) or 150 cels/mm3 blood Eos (current value) and a historical value ≥ 300 cels/mm3 or FENO ≥ 25 ppb (current value).
* Uncontrolled asthma, this is, ACT <20 and/or > 1 of an exacerbation in the last 12 months, despite treatment with ICS/LABA at medium dose.
* Written informed consent.

Exclusion Criteria:

* Patients who refuse to sign the informed consent form.
* Medical situation that prevents the collection of study information.
* Diagnosis of severe uncontrolled asthma established with criteria other than those established (ACT <20 and/or > 1 exacerbation in the last 12 months, despite treatment with ICS / LABA at medium dose).
* Medical or administrative situation that prevents the patient from following up to a minimum of 52 weeks.
* Treatment with high dose ICS/LABA, LAMA, systemic corticosteroid, azithromycin, monoclonal antibody.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
The percentage of patients controlled | At 52 weeks
  The primary endpoint will be the percentage of patients controlled at week 52, with both an ACT score of 20 or greater and no severe exacerbations.

SECONDARY OUTCOMES:
Percentage of patients controlled | At week 24
  Percentage of patients controlled at week 24, with both an ACT score of 20 or greater and no severe exacerbations.
ASMA CONTROL TEST (ACT) | At weeks 12, 24 and 52
  This is a 5-point scale. Scores range from 5 (poor asthma control) to 25 (total asthma control), with higher scores reflecting better asthma control. An ACT score >19 indicates well-controlled asthma. The minimally important difference (MID) is 3 points.
AIRQ | At weeks 12, 24 and 52
  It is a patient assessment tool intended to help identify patients aged 12 years and older whose health may be at risk due to uncontrolled asthma. It is a 10-item, equally weighted asthma control questionnaire comprising 7 impairment items and 3 risk items.
Quality of life (Mini-AQLQ) | At weeks 12, 24 and 52
  This instrument has 15 questions in the same domains as the original AQLQ (symptoms, activities, emotions and environment). A change in score greater than 0.5 can be considered clinically important.
Postbronchodilator FEV1 | At weeks 12, 24 and 52
  Performed with equipment and techniques that meet the standards developed by the Spanish Society of Respiratory Medicine (SEPAR) (18). Spirometry results will include pre-/ post-bronchodilator FEV1 (in litres) and % predicted value, FVC (in litres and % predicted) and FEV1/FVC ratio. Bronchodilator response is defined as an increase in post-bronchodilator FEV1 >12% and >0.2 l (measured 15 minutes after inhalation of 200 μg of salbutamol, using a spacer chamber) compared to pre-bronchodilator FEV1.
Severe exacerbations | At week 24 and 52
  Severe exacerbations
Differences between groups in 8 AM serum cortiso | At week 52
  Differences between groups in 8 AM serum cortiso
Adherence in the two study arms | At week 52
  Adherence in the two study arms
Factors related to triple and high-dose ICS/LABA failure and success (control) | At week 52
  Factors related to triple and high-dose ICS/LABA failure and success (control)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Pérez De Llano, MD, Principal Investigator — Sociedad Española de Neumología y Cirugía Torácica
Locations (17):
- Spain (17):
  - Hospital Universitario de A Coruña, A Coruña, A Coruña
  - Hospital General Universitario Dr. Balmis de Alicante, Alicante, Alicante
  - Hospital Comarcal de Inca - Tramuntana, Inca, Balearic Islands
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Universitario de Cruces, Barakaldo, Bizkaia
  - Hospital Universitario Galdakao-Usansolo, Galdakao, Bizkaia
  - Hospital Universitario De Jerez, Jerez de la Frontera, Cádiz
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital Universitario Clínico San Cecilio, Granada, Granada
  - Hospital Universitario Lucus Augusti, Lugo, Lugo
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Clínico Universitario de Salamanca, Salamanca, Salamanca
  - Hospital de Sagunto, Sagunto, Valencia
  - Hospital Universitario Doctor Peset, Valencia, Valencia
  - Hospital Costa del Sol, Marbella, Álaga

IPD SHARING:
Plan to Share IPD: No